CLINICAL TRIAL: NCT06409572
Title: Study of GeneXpert MTB/RIF Versus the Routine Methods for Detection of Mycobacterium Tuberculosis
Brief Title: Study of GeneXpert Mycobacterium Tuberculosis/ Rifampicin (MTB/RIF) Versus the Routine Methods for Detection of Mycobacterium Tuberculosis
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Hussien Mahran Shehata, Principal Investigator, Sohag University
Other Study IDs: Soh-Med-24-4-08MD
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: GeneXpert MTB/RIF — Rapid and accurate method for detection of tuberculosis.

SUMMARY:
1. Compare the performance of GeneXpert method with the routine methods including smear microscopy and Lowenstein-Jensen (LJ) media culture to choose the best available test for the diagnosis of TB.
2. To assess the GeneXpert MTB/RIF assay performance in detection of Mycobacterium tuberculosis in smear-negative sputum samples.

DETAILED DESCRIPTION:
Tuberculosis (TB) infection, caused by Mycobacterium tuberculosis, is a leading cause of mortality worldwide and ranks among the deadliest infectious diseases, including HIV and malaria. Despite global efforts, TB remains a significant public health threat, particularly in developing and underdeveloped countries. The World Health Organization (WHO) has reported that an estimated 10.4 million people contract new TB infections yearly, with 1.8 million TB-related deaths occurring annually.

TB usually affects the lungs, but it can also affect other parts of the body, such as the brain, spine, and many other organ systems. The most common form is pulmonary TB, which is easily spread by aerosol droplets. If another person inhales air containing these droplet nuclei, the probability of getting infected is very high. The chance of transmissibility increases if there is a delay in disease detection and treatment initiation.

Tuberculosis is an infection that requires extensive treatment. Active pulmonary TB patients can transmit the infection through the air then the droplet nuclei move through upper respiratory tract and bronchi to reach the lungs alveoli.

It is critical to treat active pulmonary TB patients as soon as possible in order to decrease the danger of infection spreading to others. The initial stage in TB diagnosis is sputum acid fast bacillus (AFB) staining, which has an advantage of having an average turnaround time (TAT) about 24 hours.

There are a number of tests available for the diagnosis of tuberculosis each having their own limitations. Conventional microscopy has low sensitivity and culture requires longer time for positivity. The commercially available automated, liquid Mycobacterium Growth Indicator tube (MGIT) culture system is time-consuming and requires specialized laboratories. On the other side, nucleic acid amplification techniques not only provide the advantage of rapidity of diagnosis but also detect even low genomic copies in various specimens and curtail the transmission of the disease.

The World Health Organization (WHO) has endorsed the implementation of GeneXpert MTB/RIF assay for national tuberculosis programs in developing countries. The GeneXpert MTB/RIF is an automated, user friendly and rapid test based on nested real-time polymerase chain reaction (PCR) assay and molecular beacon technology for MTB detection and RIF resistance.

The results are obtained within a short period of time (2 h). Moreover this technique is not prone to cross-contamination, requires minimal Biosafety facilities and has a high sensitivity in smear-negative pulmonary TB. The diagnosis of extrapulmonary tuberculosis (EPTB) is often difficult to establish, considering that number of bacteria in specimens is often very low, a collection often requires invasive procedures, and it is not easy to obtain multiple samples. In this scenario GeneXpert is a potentially useful tool for extrapulmonary specimens.

ELIGIBILITY:
Inclusion Criteria:

All suspected tuberculous patients.

Exclusion Criteria:

* children
* Previously diagnosed patients.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Sampling:Morning sputum samples or any suspected fluid as pleural or pus.
  2. Laboratory investigations:
     1. Direct Smear Preparation and Ziehl-Neelsen staining.
     2. MTB culture on Lowenstein-Jensen (LJ) media
     3. Gene-Xpert MTB/RIF assay.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Compare the performance of GeneXpert method with the routine methods including smear microscopy and Lowenstein-Jensen (LJ) media culture to choose the best available test for the diagnosis of TB. | Baseline

REFERENCES:
- [Background] AGRAWAL, M., BAJAJ, A., BHATIA, V. & DUTT, S. 2016. Comparative study of GeneXpert with ZN stain and culture in samples of suspected pulmonary tuberculosis. Journal of clinical and diagnostic research: JCDR, 10, DC09. GONG, X., HE, Y., ZHOU, K., HUA, Y. & LI, Y. 2023. Efficacy of Xpert in tuberculosis diagnosis based on various specimens: a systematic review and meta-analysis. Frontiers in Cellular and Infection Microbiology, 13, 500. GUENAOUI, K., HARIR, N., OUARDI, A., ZEGGAI, S., SELLAM, F., BEKRI, F. & TOUIL, S. C. 2016. Use of GeneXpert Mycobacterium tuberculosis/rifampicin for rapid detection of rifampicin resistant Mycobacterium tuberculosis strains of clinically suspected multi-drug resistance tuberculosis cases. Annals of translational medicine, 4. KHAN, A. S., ALI, S., KHAN, M. T., AHMED, S., KHATTAK, Y., IRFAN, M. & SAJJAD, W. 2018. Comparison of GeneXpert MTB/RIF assay and LED-FM microscopy for the diagnosis of extra pulmonary tuberculosis in Khyber Pakhtunkhwa, Pakistan. brazilian journal of microbiology, 49, 909-913. KHATER, E. S. & ABDO, K. H. 2022. Role of Gene-Xpert MTB/RIF assay in detection of Mycobacterium tuberculosis in smear-negative sputum samples. Microbes and Infectious Diseases, 3, 606-614. WILLIAM, T., PARAMESWARAN, U., LEE, W. K., YEO, T. W., ANSTEY, N. M. & RALPH, A. P. 2015. Pulmonary tuberculosis in outpatients in Sabah, Malaysia: advanced disease but low incidence of HIV co-infection. BMC infectious diseases, 15, 1-9. ZUMLA, A., GEORGE, A., SHARMA, V., HERBERT, R. H. N., OXLEY, A. & OLIVER, M. 2015. The WHO 2014 global tuberculosis report-further to go. The Lancet Global Health, 3, e10-e12.